CLINICAL TRIAL: NCT05034640
Title: Pain Versus Gain: Multiport Versus Single-Port Thoracoscopic Surgery for Pediatric Pneumothorax a Case Series
Brief Title: Single Site Thoracic Surgery for Pediatric Pneumothorax
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5210158
Record Dates: First submitted 2021-08-17; First posted 2021-09-05 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Disorder; Pneumothorax, Spontaneous; Thoracic Diseases; Thoracic Surgery
MeSH Terms: conditions — Pneumothorax; Thoracic Diseases | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Multiport Thoracoscopic Surgery for Pediatric Pneumothorax: Patients who had multiport video assisted thoracoscopic surgery for pediatric pneumothorax.
  Interventions: Procedure: Conventional multiport thoracoscopic surgery
- Single Port Thoracoscopic Surgery for Pediatric Pneumothorax: Patients who had single port video assisted thoracoscopic surgery for pediatric pneumothorax.
  Interventions: Procedure: Single port site thoracoscopic surgery

INTERVENTIONS:
Procedure: Conventional multiport thoracoscopic surgery — Use 2 or more incisions for multiple instrument entry during the surgery and chest tube placement at the end of the operation.
  Other Names: Video assisted thoracoscopic surgery, multi-incisions
  Groups: Conventional Multiport Thoracoscopic Surgery for Pediatric Pneumothorax
Procedure: Single port site thoracoscopic surgery — Using only 1 incision for multiple instrument entry during the surgery and chest tube placement at the end of the operation. Single port - GelPOINT Mini® port (Applied Medical, Rancho Santa Margarita, California, USA)
  Other Names: Single incision video assisted thoracoscopic surgery
  Groups: Single Port Thoracoscopic Surgery for Pediatric Pneumothorax

SUMMARY:
Video-Assisted Thoracoscopic Surgery (VATS) has become a standard of care in adults, pediatric surgeons have been slower to undertake this approach. There are limitations for working in children. The site of a chest tube becomes the working site for thoracoscopic surgery and the only scar. We propose this study to do a retrospective review comparing the conventional multiport thoracic surgery with the newer single port site.

DETAILED DESCRIPTION:
While Video-Assisted Thoracoscopic Surgery (VATS) has become a standard of care in adults, pediatric surgeons have been slower to undertake this approach. The limitations for working in children are decreased working space, unknown thoracoscopic effects on body physiology, and instrument accommodation. Especially as the field for minimally invasive surgery expands, using the single port approach has unique implications in children. The site of a chest tube becomes the working site for thoracoscopic surgery and the only scar. Despite some learning curve, the preliminary outcomes are similar to the multiport surgeries with better cosmesis. The learning curves for single port site surgery have been well described and our group recently performed a similar study for appendectomies. We propose this study to do a retrospective review comparing the conventional multiport thoracic surgery with the newer single port site.

ELIGIBILITY:
Inclusion Criteria:

* Age < 19 years old
* pneumothorax
* underwent surgery for pneumothorax

Exclusion Criteria:

* Age =/> 19 years old
* history of prior thoracic surgery
* history of cancer

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (age <19 years old) who presented to our hospital for the treatment of pneumothorax. Some patients were transferred from outside facilities, but did not have prior thoracic surgery or history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Total amount of opioid doses in 24 hours post-op | 24 hours post-operative VATS procedure
  Pain medication records will be reviewed for all opioids dispensed during the post-operative period until time of discharge. The name of the opioid, the dosage, the route, and the frequency will be recorded.period until time of discharge. The name of the opioid, the dosage, the route, and the frequency will be recorded.
Assessment of length of time of chest tube insertion | Time from surgery until chest tube removal
  Time will be recorded from surgery until chest tube removal post operation.

SECONDARY OUTCOMES:
Assessment of operation time | The time from surgery incision start to surgery closing will be the end time.
  The length of surgery will be recorded.
Assessment of pneumothorax reoccurrence | Within 48 hours post-operative period after surgery.
  If a pneumothorax occurs in the post-operative period, this will be recorded.
Total opioid dose from surgery until discharge | Within 72 hours post-operative period after surgery.
  Pain medication records will be reviewed for all opioids dispensed during the period from start of surgery through time of hospital discharge. The name of the opioid, the dosage, the route, and the frequency will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Radulescu, MD, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol and data will be shared amongst study staff.
Supporting Information: Study Protocol
Time Frame: The protocol will become available after the study start and for 3 years after the study completion.
Access Criteria: Pediatric surgeon, request to primary investigator.

REFERENCES:
- [Background] Fernandez-Pineda I, Seims AD, VanHouwelingen L, Abdelhafeez H, Wu H, Wu J, Murphy AJ, Davidoff AM. Modified Uniportal Video-Assisted Thoracic Surgery Versus Three-Port Approach for Lung Nodule Biopsy in Pediatric Cancer Patients. J Laparoendosc Adv Surg Tech A. 2019 Mar;29(3):409-414. doi: 10.1089/lap.2018.0120. Epub 2018 Nov 10. PMID 30418096
- [Background] Song IH, Lee SY, Lee SJ. Can single-incision thoracoscopic surgery using a wound protector be used as a first-line approach for the surgical treatment of primary spontaneous pneumothorax? A comparison with three-port video-assisted thoracoscopic surgery. Gen Thorac Cardiovasc Surg. 2015 May;63(5):284-9. doi: 10.1007/s11748-015-0522-2. Epub 2015 Jan 29. PMID 25630836
- [Background] Martynov I, Lacher M. Homemade Glove Port for Single-Incision Pediatric Endosurgery (SIPES) Appendectomy-How We Do It. European J Pediatr Surg Rep. 2018 Jan;6(1):e56-e58. doi: 10.1055/s-0038-1667140. Epub 2018 Jul 24. PMID 30046510
- [Background] Zimmermann P, Martynov I, Perger L, Scholz S, Lacher M. 20 Years of Single-Incision-Pediatric-Endoscopic-Surgery: A Survey on Opinion and Experience Among International Pediatric Endosurgery Group Members. J Laparoendosc Adv Surg Tech A. 2021 Mar;31(3):348-354. doi: 10.1089/lap.2020.0797. Epub 2020 Dec 31. PMID 33395367
- [Background] Goodman LF, Lin AC, Sacks MA, McRae JJLH, Radulescu A, Khan FA. Single site versus conventional laparoscopic appendectomy: some pain for no gain? J Surg Res. 2021 Aug;264:321-326. doi: 10.1016/j.jss.2021.03.010. Epub 2021 Apr 10. PMID 33848830